CLINICAL TRIAL: NCT02007889
Title: The Effect of L-carnitine on the Prevention of Renal Scarring in Children With Acute Pyelonephritis
Brief Title: L-carnitine on the Prevention of Renal Scarring in Acute Pyelonephritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Azadeh Eshraghi, Clinical Pharmacist, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ShahidBU
Record Dates: First submitted 2013-09-21; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Acute Pyelonephritis(APN)
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- L-carnitine (Active Comparator): 50 mg/kg/day carnitine in divided 2-3 times/day (maximum 3 g/day) in addition to antibiotic regimens
  Interventions: Drug: L-carnitine
- Control (No Intervention): control group received just antibiotic regimens without L-carnitine

INTERVENTIONS:
Drug: L-carnitine — 50 mg/kg/day carnitine in divided 2-3 times/day (maximum 3 g/day) in addition to antibiotic regimens
  Arms: L-carnitine

SUMMARY:
Risk factors for parenchymal damage in urinary tract infection are vesicoureteral reflux (VUR),obstructive uropathy,the number of flares of acute pyelonephritis(APN) and delay in treatment of acute infection.The pathogenesis of APN is related to bacterial virulenece,immune response,tissue factors,apoptosis and production of free radicals that lead to fibrosis and renal scarring. Oxidative stress in renal cells may be a critical factor in the pathogenesis of pyelonephritis whereas pharmacological management of the oxidative stress response may provide a therapeutic effect in preventing renal pathologies. Animal model show that L-carnitine alleviated oxidative stress, and acute renal inflammatory injury can be prevented much more effectively by carnitine in addition to conventional antibiotic treatment in pyelonephritis.This study is a simple randomized clinical trial (RCT) evaluating the effect of L-carnitine in addition to antibiotic on preventing renal scaring after acute pyelonephritis in children. Simple non- blind randomized clinical trial on 78 patients in 2 groups (intervention & control) is conducted.Children aged 1 month to 10 years with positive urine culture, clinical findings, and 99mTc-dimercaptosuccinic acid (DMSA) scintigraphy-based evidence in favor of acute pyelonephritis were enrolled into a clinical trial. Patients were excluded if they had neurogenic bladder, systemic hypertension, obstructive uropathy. Patients in Intervention group are administered 50 mg/kg/day carnitine in divided 2-3 times/day (maximum 3 g/day) in addition to antibiotic regimens and patients in control group received antibiotic regimens. Primary outcome is the development of renal scar by doing DMSA renal scan on the 7th day of admission and six months after the intervention and compared between groups and secondary outcome is the incidence and severity of pyelonephritis and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 10 years with positive urine culture, clinical findings, and 99mTc-dimercaptosuccinic acid (DMSA) scintigraphy-based evidence in favor of acute pyelonephritis

Exclusion Criteria:

* neurogenic bladder,
* systemic hypertension,
* obstructive uropathy

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Development of renal scar by doing DMSA renal scan | Seven and six months after the intervention

SECONDARY OUTCOMES:
Severity of pyelonephritis and response to treatment. | Six month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Golnaz Vaseghi, Ph.D pharmacology, Principal Investigator — Physiology Research Center; Alaleh Gheisari, Principal Investigator — Pediatric Nephrologist,Isfahan University, Isfahan, Iran; Nahid Aslani, Resident of pediatrics, Principal Investigator — Isfahan University of Medical Sciences; Azadeh Eshraghi, Clinical Pharmacist, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences,Alzahra Hospital, Isfahan, Isfahan, Iran